CLINICAL TRIAL: NCT05383651
Title: International Prospective Multicenter Observational Study of the Safety and Performance of Bellavista Ventilator and the IFLow Sensor During Routine Use in the Neonatal, Pediatric, and Adult Intensive Care Unit
Brief Title: Post Market, Prospective Multicenter Observational Study of the Safety and Performance of Bellavista Ventilator
Status: Completed | Type: Observational
Sponsor: Vyaire Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: 100-P0243
Record Dates: First submitted 2022-04-21; First posted 2022-05-20 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Ventilation Therapy; Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Adults
  Interventions: Device: bellavista 1000
- Pediatric/ Neonates
  Interventions: Device: bellavista 1000 neo

INTERVENTIONS:
Device: bellavista 1000 — observational use of Bellavista 1000 ventilator in adult ventilated patients
  Groups: Adults
Device: bellavista 1000 neo — observational use of Bellavista 1000 ventilator in neonatal ventilated patients
  Groups: Pediatric/ Neonates

SUMMARY:
This prospective post market clinical follow up (PMCF) study will evaluate the safety and performance of bellavista ventilator and the iFlow sensors in daily clinical routine.

DETAILED DESCRIPTION:
A prospective, multicenter, single-cohort post market observational study, which will analyze data from neonatal, pediatric and adult patients, who are ventilated with the bellavista ventilator.

Ventilator data are continuously recorded in the bellavista ventilator. Patient related data will be recorded in an electronic case report form (CRF). Data from the ventilator and the eCRF are then combined and the primary and secondary endpoints calculated.

ELIGIBILITY:
Inclusion Criteria:

* Patient ventilated with bellavista
* Patient in ICU setting
* Signed informed consent per ethical committee requirements

Exclusion Criteria:

* Patients expected to be ventilated less than 12 hours
* The clinical care team does not agree with inclusion of the patient to the study

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Neonates and adults ventilated with Bellavista ventilator in intensive care units.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Ventilator Performance - Relationship between the set and observed Positive End-Expiratory Pressure (PEEP) | through study completion, an average of 12 hours- 24 days
  Difference between set and observed PEEP
Ventilator Performance - Relationship between the set and observed Peak Inspiratory Pressure (PIP) | through study completion, an average of 12 hours- 24 days
  Difference between set and observed PIP
Ventilator Performance - Relationship between the set and observed Continuous Positive Airway Pressure (CPAP) | through study completion, an average of 12 hours- 24 days
  Difference between set and observed CPAP
Ventilator Performance - Relationship between the set and observed tidal volume | through study completion, an average of 12 hours- 24 days
  Difference between set and observed tidal volume
Ventilator Performance - Relationship between the set and observed flow rate | through study completion, an average of 12 hours- 24 days
  Difference between set and observed flow rate

SECONDARY OUTCOMES:
Ventilator Safety - Device failure rate | through study completion, an average of 12 hours- 24 days
  malfunction of the ventilators necessitating removal of a patient to another ventilation mode or ventilator (bellavista technical alarms with ID higher than 300)
Ventilator Safety - Descriptive statistical analysis of all ventilator alarm events | through study completion, an average of 12 hours- 24 days
  A summary table presenting number, type and duration of ventilator alarms within study population
Analysis of patient-ventilator interactions - Duration of mechanical ventilation | through study completion, an average of 12 hours- 24 days
  Number of days under invasive mechanical ventilation
Analysis of patient-ventilator interactions - Reintubation rate | through study completion, an average of 12 hours- 24 days
  Number of patients with the need of reintubation, considered by the physician in charge of the patients, after a scheduled or unplanned extubation
Length of ICU stay | through study completion, an average of 12 hours- 24 days
  Period of time that the bellavista-ventilated patients spend in the ICU before being discharged (alive or died)
Length of hospital stay | through study completion, an average of 12 hours- 24 days
  Period of time that the bellavista-ventilated patients spend in the hospital after ICU discharge
Ventilator Safety - Number of study participants with device related adverse events | through study completion, an average of 12 hours- 24 days
  Number of malfunction of the investigational device leading to potential or actual patient harm
Extubation failure | through study completion, an average of 12 hours- 24 days
  Defined as the need of reintubation within the first 48 hours from a scheduled extubation
Hospital mortality | through study completion, an average of 12 hours- 24 days
  Number of bellavista-ventilated patients who died during the hospital admission after the ICU discharge
Failure of noninvasive treatment | through study completion, an average of 12 hours- 24 days
  Need of orotracheal intubation in bellavista-ventilated patients after an attempt of noninvasive treatment (NIV and HFOT) that failed, defined by the physician in charge of the patient.
Analysis of patient-ventilator interactions - Pneumothorax rate | through study completion, an average of 12 hours- 24 days
  Number of confirmed pneumothoraxes during ventilation
Analysis of patient-ventilator interactions - Sepsis | through study completion, an average of 12 hours- 24 days
  Number of patients with sepsis
Analysis of patient-ventilator interactions - Bronchopulmonary dysplasia | through study completion, an average of 12 hours- 24 days
  Need of oxygen or positive airway pressure at 36 weeks corrected age
Analysis of patient-ventilator interactions - Retinopathy of prematurity | through study completion, an average of 12 hours- 24 days
  Number of patients with retinopathy of prematurity and level
Analysis of patient-ventilator interactions - Necrotizing enterocolitis | through study completion, an average of 12 hours- 24 days
  Number of patients with necrotizing enterocolitis
Intraventricular hemorrhage | through study completion, an average of 12 hours- 24 days
  Number of patients with intraventricular hemorrhage

CONTACTS AND LOCATIONS:
Locations (2):
- University Health Network, Toronto, Ontario, Canada
- University Children's Hospital Zürich, Zurich, Canton of Zurich, Switzerland